CLINICAL TRIAL: NCT06079216
Title: Making Connections Thru Music: A Group Music Therapy-Based Intervention for Persons With Dementia
Brief Title: Making Connections Thru Music
Acronym: MCTM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopeful Aging (Industry)
Collaborators: Benjamin Rose Institute on Aging (Other)
Responsible Party: Principal Investigator, Gregg Gorzelle, Associate Director of Research, Hopeful Aging
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HearthstoneI
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Dementia; Alzheimer Disease; Vascular Dementia
MeSH Terms: conditions — Dementia; Alzheimer Disease; Dementia, Vascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCTM Intervention (Experimental): Activity sessions will be led by activity volunteers
  Interventions: Behavioral: Volunteer Led Making Connections Thru Music
- Control (Active Comparator): Activity sessions will be led by activity professionals
  Interventions: Behavioral: Staff Led Making Connections Thru Music

INTERVENTIONS:
Behavioral: Volunteer Led Making Connections Thru Music — Volunteer led Group music therapy-based intervention
  Arms: MCTM Intervention
Behavioral: Staff Led Making Connections Thru Music — Staff led Group music therapy-based intervention
  Arms: Control

SUMMARY:
Healthcare systems around the world, including within the United States, have long-established shortages of trained caregivers. The American Health Care Association states that "the health care system has experienced a shortage of trained caregivers for critical roles for some time." This scarcity directly impacts the 45,800 Long-Term Care (LTC) communities throughout the U.S.

Concurrent with this staff shortage, more than half of LTC residents have some form of dementia. These two issues create a serious public health concern, since dementia is associated with a variety of behavioral expressions, such as aggression, anxiety, and agitation. Behavioral expressions of dementia can be successfully managed with the use of tailored, psychosocial interventions and communication support. Unfortunately, existing staff shortages make the facilitation of such interventions challenging.

One powerful and often-overlooked approach to ameliorating staffing shortages involves the utilization of retired volunteers to facilitate interventions for persons with dementia (PWD). Based on the nearly universal love of music and a promising pilot study, the product to be developed and tested in this STTR will build upon the combined prior work of the Principal Investigators. Making Connections Thru Music (MCTM), an urgently needed product, will enable retired volunteers to facilitate an evidence-based music and discussion intervention with PWD. MCTM aims to improve engagement, enhance quality of life, and reduce behavioral expressions in PWD. The intervention will consist of two main components: (1) a comprehensive online training course for volunteers, which will provide a general overview of dementia, demonstrate effective communication strategies to use with PWD, and instruct volunteers to effectively facilitate MCTM sessions, and (2) an app containing a structured MCTM intervention protocol and toolkit, which will be the means by which volunteers facilitate MCTM. MCTM will be marketed to LTC communities.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be aged 55+ and speak/read conversational English.
* Staff participants must be at least 18 years old, work within a residential care facility participating in the study, and speak and read English.

Exclusion Criteria:

* Volunteers will be excluded if they are diagnosed with dementia based on self-report and/or if they score 23 or lower on theMini Mental State Exam (MMSE; Folstein et al., 1975). Such a score would be indicative of possible cognitive impairment.
* Staff members will be excluded if they work third shift only. PWD Residents with dementia must be diagnosed with dementia (any type), score 10 or above on the MMSE, be aged 65+, and speak/read conversational English.
* PWD will be excluded if they show signs of rapid physical or cognitive decline (based upon staff report or as evidenced by information gained during screening).

Ages: 18 Years to 103 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Menorah Park Engagement Scale | Baseline (weeks 1-4) Treatment (weeks 5-12)
  The MPES is an observational scale that measures four types of engagement: Constructive Engagement, Passive Engagement, Distracted Engagement, and Non-Engagement / Apathy The MPES also measures Pleasure, defined as clearly observable smiling or laughing. For each item, the minimum possible value is 0 (not at all) and the maximum possible value is 2 (more than half of the time). For Constructive Engagement, Passive Engagement, and Pleasure, higher scores would represent a better outcome. For Distracted Engagement and Non-Engagement, higher scores would represent a worse outcome.

SECONDARY OUTCOMES:
Alzheimer's Disease Knowledge Scale | Baseline (weeks 1-4) Treatment (weeks 5-12)
  30-item scale to measure knowledge of Alzheimer's Disease. The range of score is zero to 30. A higher score indicates a better outcome.
Geriatric Depression Scale- Short Form. Scores can range from zero to 15. Higher scores suggest a worse outcome | Baseline (weeks 1-4) Treatment (weeks 5-12)
  This is a 15-item measure of depression in older adults that is conducted via direct interview.
Neuropsychiatric Inventory - Nursing Home. | Baseline (weeks 1-4) Treatment (weeks 5-12)
  The Neuropsychiatric Inventory-Nursing Home is a comprehensive assessment of psychopathology in persons with dementia, focused on people residing in nursing homes. Researchers typically use the frequency x severity (FxS) total score on this measure. We will be using this score in this study. The FxS score ranges from 0 to 120, with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hearthstone Institute, LLC, Winchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided